CLINICAL TRIAL: NCT04167202
Title: Hydrotherapy With Hydrogen-rich Water Compared With RICE Protocol Following Acute Ankle Sprain in Professional Athletes: a Randomized Non-inferiority Trial
Brief Title: Hydrotherapy With Hydrogen-rich Water vs. RICE Protocol Following Acute Ankle Sprain
Acronym: HRWAAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-HRW/2019
Record Dates: First submitted 2019-11-11; First posted 2019-11-18 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen-rich water (Experimental): Six 30-min ankle baths with hydrogen-rich water (one hydrotherapy every 4 hours)
  Interventions: Procedure: Hydrogen-rich water
- RICE protocol for acute injury (Active Comparator): RICE protocol include: (1) rest, (2) ice packs every 20 min every 3 hours (total of 8 sessions), (3) compression with elastic bandage for 24 h, and (4) leg elevation at all possible times of the injured area above the level of the heart
  Interventions: Procedure: RICE

INTERVENTIONS:
Procedure: Hydrogen-rich water — Hydrogen-rich water (one hydrotherapy every 4 hours)
  Arms: Hydrogen-rich water
Procedure: RICE — RICE protocol
  Arms: RICE protocol for acute injury

SUMMARY:
The traditional treatment of soft tissue injuries consists of the RICE protocol - rest, ice, compression, and elevation, followed for up to 72 hours after a trauma. Although designed as an immediate therapy to reduce inflammation that occurs after an acute injury, the RICE might not be the best way to promote healing due to limiting blood flow. Molecular hydrogen (H2) has recently been put forward as a possible adjuvant treatment in musculoskeletal medicine, yet limited data are available concerning its effectiveness as a first-aid intervention.

DETAILED DESCRIPTION:
Experimental protocol

* Randomized controlled parallel-group trial
* Acute (24 h) post-injury intervention:

  * Hydrogen-rich water hydrotherapy
  * RICE protocol
* First sessions given immediately after an initial examination (~ 60 min after the injury).
* Source of hydrogen-rich water = HRW Natural Health Products Inc. (New Westminster, BC, Canada)

  o Formulation (7g/ tablets, 800mg Magnesium) dissolved into a 3-L stationary whirlpool with water (20°C)
* No other interventions during the period of evaluation

Outcomes assessed at baseline (pre-intervention) and at 24-h follow up:

* Figure-of-eight method of measuring ankle joint swelling
* Visual analogue score (VAS) score for pain at rest and during movement
* Weight-bearing lunge test (WBLT)
* Single leg balance test (SLBT) with eyes open and closed
* Serum inflammatory biomarkers (IL-1ß, TNF-α, CRP) • Early termination criteria: serious subjective side effects (e.g. tingling, discoloration of skin, burning, itching, rash)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 35 years
* Body mass index 19 - 25 kg/m2
* Free of major chronic diseases or acute disorders
* Acute ankle sprain incurred during sport-related activity

Exclusion Criteria:

* History of a previous ankle sprain during the past 6 months
* Unwillingness to return for follow-up analysis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Change in ankle circumference for joint swelling | Baseline vs. 24 hours post-intervention
  Baseline vs. 24

SECONDARY OUTCOMES:
Change in VAS score for pain (0-10), higher score means worse outcome | Baseline vs. 24 hours post-intervention
  Baseline vs. 24 h

OTHER OUTCOMES:
Change in ankle mobility for maximal dorsiflexion in centimeters, higher score means worse outcome | Baseline vs. 24 hours post-intervention
  Baseline vs. 24 h
Change in single-leg balance in seconds, higher score means better outcome | Baseline vs. 24 hours post-intervention
  Baseline vs. 24 h
Change in serum levels of C-reactive protein | Baseline vs. 24 hours post-intervention
  Baseline vs. 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Nebojsa Maksimovic, PhD, Study Chair — Faculty of Sport and PE
Locations (1):
- Applied Bioenergetics Lab at Faculty of Sport and PE, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostojic SM, Vukomanovic B, Calleja-Gonzalez J, Hoffman JR. Effectiveness of oral and topical hydrogen for sports-related soft tissue injuries. Postgrad Med. 2014 Sep;126(5):187-95. doi: 10.3810/pgm.2014.09.2813. PMID 25295663
- [Background] Cole AR, Perry DA, Raza A, Nedder AP, Pollack E, Regan WL, van den Bosch SJ, Polizzotti BD, Yang E, Davila D, Afacan O, Warfield SK, Ou Y, Sefton B, Everett AD, Neil JJ, Lidov HGW, Mayer JE, Kheir JN. Perioperatively Inhaled Hydrogen Gas Diminishes Neurologic Injury Following Experimental Circulatory Arrest in Swine. JACC Basic Transl Sci. 2019 Mar 27;4(2):176-187. doi: 10.1016/j.jacbts.2018.11.006. eCollection 2019 Apr. PMID 31061920
- [Background] Ostojic SM. Should hydrogen therapy be included in a musculoskeletal medicine routine? F1000Res. 2016 Nov 10;5:2659. doi: 10.12688/f1000research.9758.1. eCollection 2016. PMID 28003879